CLINICAL TRIAL: NCT05436054
Title: A Randomised Controlled Trial to Compare Efficacy and Tolerability of Plenvu® and Picoprep® as Cleansing Agents Before Colonoscopy
Brief Title: A Trial to Compare Efficacy and Tolerability of Plenvu® and Picoprep® as Cleansing Agents Before Colonoscopy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Regionshospital Nordjylland (Other Government); Norgine (Industry)
Responsible Party: Principal Investigator, Hayder Mahmood Waheeb Alqaisi, Resident doctor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122021
Record Dates: First submitted 2022-06-20; First posted 2022-06-28 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Colon Disease
Keywords: colonoscopy; bowel cleansing
MeSH Terms: conditions — Colonic Diseases | interventions — picosulfate sodium; Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: This is a single-center, single-blinded, randomised equivalence trial to compare the efficacy and tolerability of Picoprep® and Plenvu® as cleansing agents before colonoscopy. The trial is to be performed on patients referred to Frederikshan endoscopy center for a colonoscopy, most of these patients are referred to exclude/diagnose colon cancer. Colonoscopies are performed in Frederikshavn local hospital/North Jutland/Denmark by different colonoscopists.
Who Masked: Outcomes Assessor
Masking Description: This is a single-blinded trial. The colonoscopist who performs the procedure and evaluates the quality of cleansing is blinded to which preparation was used. This is achieved during randomisation of the patient where they receive a paper form prescription, thus the colonoscopist cannot check that in the electronic system.
  Blinding is not done to the patients as the bias is considered small. Cleansing agents are not normally used in the general population and the effect of previous experience to evaluate the tolerability in the present time is not considered to be large.
  Subjects will be well informed in the participation information and in the meeting not to reveal the type of cleansing they received to the colonoscopist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Picoprep (Active Comparator): Picoprep®:
  Active substances: An envelope Picoprep® contains 10 mg sodium picosulfate, 3,5 g magnesium oxide, and 12 g citric acid.
  Mechanism of action: Sodium picosulfate is a peristaltic agent that increases the peristalsis of the intestine. Magnesium oxide and citric acid are osmotic agents to increase water content in the bowel.
  Dosage and administration: consist of 2 envelopes, the first envelope, after dissolving in 150 ml water, should be taken 10-18 hours before the colonoscopy, then at least 250mlX5 clear fluid (not only water) over the next hours before the second dose is taken. The second envelope should be taken 4-6 hours before colonoscopy followed by 250mlX3 clear fluid (not only water) over the next hours before colonoscopy. The total fluid intake is approximately 2.3 L.
  Interventions: Drug: Picoprep
- Plenvu (Experimental): Plenvu®:
  Active substances:
  Dose nr. 1
  1 envelope contains 1 g potassium chloride, 100 g macrogol 3350, 2 g sodium chloride, and 9 g sodium sulfate.
  Dose nr. 2 1 envelope A contains 1,2 g potassium chloride, 40 g macrogol 3350, and 3,2 g sodium chloride.
  1 envelope B contains 7,54 g ascorbic acid (Vit. C) and 48,11 g sodium ascorbate.
  Mechanism of action: Macrogol 3350 is an osmotic laxative. The added electrolytes are to prevent electrolyte shifting and systemic disturbances.
  Dosage and administration: two separate nonidentical 500 ml doses are given. 2-day regime: dose nr.1 envelope is dissolved in 500 ml post water and drunk over 30 minutes. Should be taken at 6 o'clock evening before colonoscopy day. Dose nr.2 envelope A and B are dissolved in 500 ml post water and drunk over 30 minutes. Should be taken at 6 o'clock on the morning of colonoscopy day.
  After each dose of the dissolved Plenvu®, the patient should drink at least 500ml clear fluid.
  Interventions: Drug: Plenvu

INTERVENTIONS:
Drug: Picoprep — 200 patients will be randomised to this arm
  Arms: Picoprep
Drug: Plenvu — 200 patients will be randomised to this arm
  Arms: Plenvu

SUMMARY:
The trial is about comparing the efficacy of Plenvu with Picoprep. Both are bowel cleansing agents prior to visual examination of the large bowel to exclude cancer disease.

400 patients who are referred for colonoscopy to a single center in North Jutland will be randomised either to Picoprep or Plenvu. These patients will then answer a questionnaire prior to colonoscopy. The questionnaire is about the most common expected side effects and the experience of cleansing og intake of the bowel agents.

The effect of the two agents will examined using a special scoring system (Harefield) to determine the quality of bowel cleansing. Colonoscopist who evaluate the cleansing is blinded to which agent the patient has taken.

DETAILED DESCRIPTION:
Abbreviations:

PEG: Polyethelynglycol PEG-ELS: Polyethelynglycol-electrolytes lavage solution SPMC: Sodium picosulfate/magnesium citrate L: liter ex.: example Ml: milliliter eGFR: estimated glomerular filtration rate G: gram WHO - World Health Organization CIOMS - Council of International Organizations of Medical Sciences ICH - International Conference on Harmonisation

Introduction:

1. Aim of the study:

   The study aims to compare the efficacy and tolerability of the relatively new bowel preparation Plenvu® with the well-established bowel preparation Picoprep® as cleansing agents before colonoscopy. This is to test whether the low volume PEG-ELS preparation Plenvu® would have non-inferior efficacy on bowel cleansing compared with Picoprep® with a comparable effect on compliance and tolerability.
2. Background Colonoscopy is one of the most performed procedures around the world, both for diagnostic and therapeutic purposes. The number of colonoscopies in Denmark has markedly risen after the national program for colorectal cancer screening was started in 2014. Only for screening purposes, 23.532 colonoscopies were performed in 2019 .

   Adequate bowel preparation before a colonoscopy is critical for adequate colonic mucosa assessment. Poor preparation reduces the detection rate of colonic lesions and results in 10-20 % of colonoscopies failure . Many factors have been associated with inadequate bowel preparation, including failure to follow preparation instructions, and primary reasons given for this noncompliance included patient discomfort or, in the case of PEG preparations, an inability to ingest the required fluid volume. Adequate tolerability to bowel preparation and compliance with the intake of the cleansing agents will therefore lead to better preparation and a better colonoscopy success rate. Generally, the choice of cleansing agents should depend on the efficacy, tolerability, cost, and patient-related factors ( contraindications to some of the agents).

   The most commonly used preparations for bowel cleansing in Denmark are isotonic preparations like PEG-ELS (Polyethelynglycol-electrolytes lavage solution) (ex. Moviprep®, Plenvu®), and a combination preparation of both stimulant (Sodium picosulphate) and osmotic (Citric acid) laxatives (ex. Picoprep®) PEG-based preparation is known for its demand to drink a large amount of fluid. On the other hand Sodium picosulphate, based preparation is known for its relatively low safety margin and limitation of use in patients with renal/heart insufficiency, especially in old age due to the risk of electrolyte disturbance. This is possibly an issue in screening patients, especially old age because a possible underlying heart or kidney disease in a screening patient is not expected to be known by the secretary of the regional coordination centers (in Denmark) who are responsible for inviting and preparing those patients for colonoscopy.

   A meta-analysis comparing PEG to Sodiumpicosulphate/magnesium-citrate as bowel cleansing agents shows the non-inferiority of the latter in efficacy with a better adverse events profile, it shows as well a higher proportion of patients were likely to complete SPMC preparation (RR 1.08; 95 % CI 1.04-1.13, P < 0.001) and were willing to repeat it.

   A very low volume 1 L PEG-based bowel cleansing preparation (Plenvu®) was introduced recently. A multi-center observational study that compared it with low volume 2L PEG-based preparation (Moviprep®) and a conventional volume 4 L PEG preparation (Selgesse®) and the results were in favor of 1 L preparation in terms of tolerability with comparable efficacy.

   The head-to-head comparison of very low volume PEG preparation with sodium picosulfate based preparation is sparse in the literature.

   Therefore investigators aim to compare the two preparation in terms of efficacy and tolerability, and the results would be suitable for use as a basis for decision in the endoscopy centers when it comes to the choice of the cleansing preparation in the future.
3. Cleansing agents to be tested:

Both agents are approved for medical use in Denmark and are intended (in this trial) to be used in their approved indications (cleansing agents prior to Colonoscopy)

Picoprep®:

Active substances: An envelope Picoprep® contains 10 mg sodium picosulfate, 3,5 g magnesium oxide, and 12 g citric acid.

Mechanism of action: Sodium picosulfate is a peristaltic agent that increases the peristalsis of the intestine. Magnesium oxide and citric acid are osmotic agents to increase water content in the bowel.

Dosage and administration: consist of 2 envelopes, the first envelope, after dissolving in 150 ml water, should be taken 10-18 hours before the colonoscopy, then at least 250mlX5 clear fluid (not only water) over the next hours before the second dose is taken. The second envelope should be taken 4-6 hours before colonoscopy followed by 250mlX3 clear fluid (not only water) over the next hours before colonoscopy. The total fluid intake is approximately 2.3 L.

Contraindications: severe renal failure (eGFR<30), rhabdomyolysis, heart failure, hypermagnesemia, severe dehydration, Intestinal obstruction, inflammatory bowel disease, bowel perforation, and gastric retention Side effects: The most common side effects are headache, abdominal pain, nausea and vomiting, and risk for electrolytes disturbances. (Detailed description of side effects in the attached product resumé)

Plenvu®:

Active substances:

Dose nr. 1

1 envelope contains 1 g potassium chloride, 100 g macrogol 3350, 2 g sodium chloride, and 9 g sodium sulfate.

Dose nr. 2 1 envelope A contains 1,2 g potassium chloride, 40 g macrogol 3350, and 3,2 g sodium chloride.

1 envelope B contains 7,54 g ascorbic acid (Vit. C) and 48,11 g sodium ascorbate.

Mechanism of action: Macrogol 3350 is an osmotic laxative that increases water retention in the bowel and makes feces soft. The added electrolytes are to prevent electrolyte shifting and systemic disturbances.

Dosage and administration: two separate nonidentical 500 ml doses are given either in a 2-day or single-day regime. In this trial, we're using the 2-day regime.

2-day regime: dose nr.1 envelope is dissolved in 500 ml post water and drunk over 30 minutes. Should be taken at 6 o'clock evening before colonoscopy day. Dose nr.2 envelope A and B are dissolved in 500 ml post water and drunk over 30 minutes. Should be taken at 6 o'clock on the morning of colonoscopy day.

After each dose of the dissolved Plenvu®, the patient should drink at least 500ml clear fluid. Thus a total of 2L fluid at the end of preparation.

Side effects: The most common side effects are abdominal pain, nausea, body temperature rising, and anal irritation.

Contraindications: Intestinal obstruction, inflammatory bowel disease, bowel perforation, gastric retention, G6PD Caution: with severe renal failure (eGFR <30), electrolytes and fluid balance should be monitored.

With both preparations, the patient should not eat seed-containing food 5 days before the colonoscopy day. The day before the procedure only fluid diet (all that can run through a sieve) until 6 hours before the procedure and then clear fluids up to two hours before the procedure.

Trial design:

This is a single-center, single-blinded, randomised equivalence trial to compare the efficacy and tolerability of Picoprep® and Plenvu® as cleansing agents before colonoscopy. The trial is to be performed on patients referred to Frederikshan endoscopy center for a colonoscopy, most of these patients are referred to exclude/diagnose colon cancer. Colonoscopies are performed in Frederikshavn local hospital/North Jutland/Denmark by different colonoscopists.

Blinding:

This is a single-blinded trial. The colonoscopist who performs the procedure and evaluates the quality of cleansing is blinded to which preparation was used. This is achieved during randomisation of the patient where they receive a paper form prescription, thus the colonoscopist cannot check that in the electronic system.

Blinding is not done to the patients as the bias is considered small. Cleansing agents are not normally used in the general population and the effect of previous experience to evaluate the tolerability in the present time is not considered to be large.

Subjects will be well informed in the participation information and in the meeting not to reveal the type of cleansing they received to the colonoscopist.

5.2.2 Randomisation: Randomisation is conducted after the patient has signed the informed consent. Randomisation is taken in 20 blocks and each block with 20 patients(block-randomisation), using approved statistical software e.g. RedCap with help from a statistician The patient gets a trial number according to the software where each patient is randomised to either Plenvu or Picoprep. This number will be used on the questionnaire and The Harefield cleansing scale. None of the above is expected to reveal blinding for the colonoscopist.

3 Method: Patients who are referred for a colonoscopy for diagnostic/therapeutic indications (mostly to exclude cancer) are first (as a standard procedure to all patients referred for colonoscopy to Frederikshavn center) controlled by a consultant doctor (and in this trial one of the main investigators) for the indication of colonoscopy and their general conditions, at this point through out the referral letter and the patient journal the inclusion/exclusion criteria are controlled. These information would include personal, contact, health status and medical list information. These information will be passed on from the treating doctor to the main investigator . Informations will be uses to evaluate the potential subject for the inclusion and exclusion criteria and to recruit the them, and this would happen before the patient has given consent. The patient can first be contacted after confirmation from the treating doctor. This is in concordance with "Sundhedslovens § 46, stk. 1" The patient is then contacted by the secretary by telephone and the sole purpose of this contact is to tell the patient about the possibility to send the participation information and general information about the trial is given. If the patient is interested to participate in the trial the secretary will send the patient in their safe mailbox detailed information about the study (participation information), and written informed consent.

The patient is offered a detailed meeting either by a physical meeting or by telephone (its is up to the patient to choose) to be informed thoroughly about the trial. The meeting would be performed by a delegated nurse and if needed by one of the investigators. The patient is informed both by telephone and in the written information document about the meeting which would be hold in a specific time during official working hours in Frederiishavn center, are also informed about the right to a legal representative or an assistant that can attend the meeting (the patient is responsible for arranging that). After the patient has been to the meeting he/she have the right to 1 days reflection time from the meeting, if they don't respond within the period, they would be dropped from the trial and treated as usual. When the patient agrees to the terms of participation after the meeting and the reflection time they sign the informed consent either during the meeting or electronically using (NemID), if they wanted to use their reflection time. The consent is also to be signed by one of the responsible investigators (as to confirm that the patient has received all the necessary information).these patients are then randomised either to Plenvu® or Picoprep®. Prescription of the randomised preparation, instructions of intake, and general information about the procedure (Colonoscopy) are then sent to the patient in their mailbox.

Note: the reflection time can not be longer due to the fact that all patients referred for colonoscopy to exclude cancer should get their colonoscopy within 2 weeks and longer reflection time would potentially delay the process.The Cleansing agents are retrieved from any pharmacy and the bill is paid by the Region of North Jutland. That is to say that subjects participating in this trial receive the medications free of charge. This is as well the reason why no drug accountability logs will be made in this study. There is no need for dispensation for delivering medicine free of charge in concordance with BEK nr. 695 af 12. juni 2013, §13.

The patients will receive in their e-boks, while they receive the prescription for the cleansing agent, a document that declares the medicine they are receiving is a trial medicine. The document will contain the trial identification number (EudraCT. Number) and contact information for the investigator (Name, telefon number and work address)

Harefield Cleansing Scale:

When the procedure is done, the colonoscopist grades bowel preparation according to Harefield Cleansing Scale. The cleansing quality is measured after dividing the colon into 5 segments (Rectum, sigmoid colon, Descending colon, Transverse colon, and Ascending colon/Cecum) and each segment is scored from 0 (irremovable heavy hard stool), 1 (Semi-solid, only partially removable stools), 2 (Brown liquid/removable semi-solid stools) 3 (Clear liquid), and 4 (empty and clean), then a total grade is given. Grade A (all segments scored 3 or 4) and B (one or more segments scored 2) are considered as successful cleansing. Grade C (one or more segments scored 1) and D (one or more segments scored 0) is considered unsuccessful cleansing.

Canceled colonoscopies because of bad preparation will be included in the final results, and these patients will be invited to a new colonoscopy with the use of usual cleansing bowel agents (these patients are excluded from randomisation in the study again).

Tolerability questionnaire:

When the patient meets to the planned procedure, he/she receives a tolerability questionnaire to be answered before the procedure is done. This is to measure the general tolerability of the patients to the two bowel agents during the preparation period by measuring the ability to drink the whole preparation and the onset of some of the common side effects. A previously validated tolerability questionnaire is used to measure this, the original questionnaire is in English. Following changes were taken to the original questionnaire: Addition of a single question regarding the total amount of fluid the patient was able to drink as a percentage of the total required fluid was taken, and the visual assisted score testing the general tolerability is changed to a numeric score from 0 to 10. The questionnaire is translated from English to Danish and then retranslated from Danish to English by a non-healthcare-related person then the two English versions were compared to ensure validation of the Danish translation This questionnaire contains questions about the most common side effects (occurs between 10 to 1%) for both Plenvu® and Picoprep®, this would make it possible to register these in our trial.

It will as will draw a general picture about how the subjects experienced the cleansing process.

The expected duration of patient participation in the study and follow-up:

Patients are enrolled after meeting the inclusion/exclusion criteria and signing the written consent and terminated after 30 hours from ingesting the last dose of the cleansing agent.

Rules for termination of the trial:

The trial is terminated when a sample of 400 subjects has participated in the study.

Data management:

The study will be submitted to the Northern Region of Denmark ("Forskningsanmeldelse Region Nordjylland - Registrering af forskningsprojekter"). Standard operating procedures (SOPs) for data handling and record-keeping exist within the research center and these will be followed.

Data recording in form of questionnaires and bowel cleansing assessment forms will be filled when a participant has been to the procedure and Any corrections will be made in such a way that information from the original version is still available. The changes are endorsed by initials and date. All forms are filled out during (or immediately after) the assessment of a participant.

Hardcopies of data will be stored in the corresponding center and rules of personal data protection will be respected.

Electronic case report forms:

REDCap, a secure browser-based software, will be used for filling in the eCRF form for each participant. REDCap meets all regulatory safety requirements and is approved for data collection by the North Jutland Region in Denmark.

Data related to the primary and secondary outcome will be entered directly into electronic CRFs using REDCap, licensed by Aalborg University Hospital, and saved electronically. Errors and corrections are logged as provided by the REDCap interface. It is possible to export validated data from REDCap to another statistical program (e.g. SPSS) for further statistical analysis. When data have been entered, reviewed, and verified the data will be frozen to prevent editing. Digitalized data are backed up and stored on specific drives at each site under the responsibility of the investigators.

Source data identification and protection A Patient Identification List containing patient numbers, full name, civil registration number for all participants included in the study is created, and ethics according to "databeskyttelsesforordningen" and "databeskyttelsesloven" is ensured. The list is populated and updated by a project secretary or other delegated persons. All source documentation will be stored on a secure drive under the responsibility of the investigator.

Statistics and analysis:

1. Analysis The primary endpoint which is measuring efficacy using the Harefield score would classify the patient as a satisfactory and not satisfactory cleansing process. This would make analysis feasible using two by two table and Chi-Square and a p-value of less than 0.05 would be considered significant.

   The confidence interval is 95% Null hypothesis: Plenvu is not inferior to Picoprep regarding efficacy. The secondary endpoint would be described using qualitative descriptive measures.
2. Sample size The sample size is power calculated to be 400 patients using the Slovin's Formula assuming the population size is the Danish population (approximately 5,9 million) and the margin of error is 0.05.

It is computed as n = N / (1+Ne2). whereas: n = no. of samples N = total population e = error margin / margin of error The margin of error is chosen to be 0.05 as investigator choose a confidence interval of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant colonoscopy
* Older than18

Exclusion Criteria:

* Younger than 18
* Known with severe heart failure
* Known with severe renal failure (eGFR<30)
* Known for colonic stenosis
* Pregnant or breastfeeding
* Acute colonoscopy
* Cancer screening program colonoscopy
* Mentally retarded
* Redo colonoscopy of patients included in this study and colonoscopy was canceled because of bad bowel preparation.
* Patients with Phenylketonuria
* Patients with Glucose-6-phosphate-dehydrogenase deficiency
* Patients with colon or rectum resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of cleansing agent | 18 hours
  The primary endpoint is the efficacy of cleansing preparations measured by the quality of cleansing. This is done using the validated Harefield Cleansing Scale.
  The cleansing quality is measured after dividing the colon into 5 segments (Rectum, sigmoid colon, Descending colon, Transverse colon, and Ascending colon/Cecum) and each segment is scored from 0 (irremovable heavy hard stool), 1 (Semi-solid, only partially removable stools), 2 (Brown liquid/removable semi-solid stools) 3 (Clear liquid), and 4 (empty and clean), then a total grade is given. Grade A (all segments scored 3 or 4) and B (one or more segments scored 2) are considered as successful cleansing. Grade C (one or more segments scored 1) and D (one or more segments scored 0) is considered unsuccessful cleansing.

SECONDARY OUTCOMES:
Tolerability to the cleansing agent | 18 hours
  The secondary endpoint is the tolerability of the patient to cleansing preparation. This is measured using a previously validated tolerability questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Andersen, Consultant, Study Director — Region of North Jutland
Locations (1):
- Aalborg University hospital, Aalborg, North Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cash BD, Moncrief MBC, Epstein MS, Poppers DM. Patient experience with NER1006 as a bowel preparation for colonoscopy: a prospective, multicenter US survey. BMC Gastroenterol. 2021 Feb 15;21(1):70. doi: 10.1186/s12876-021-01605-y. PMID 33588763
- [Background] Byrne MF. The curse of poor bowel preparation for colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1587-90. doi: 10.1111/j.1572-0241.2002.05855.x. No abstract available. PMID 12135005
- [Background] Ness RM, Manam R, Hoen H, Chalasani N. Predictors of inadequate bowel preparation for colonoscopy. Am J Gastroenterol. 2001 Jun;96(6):1797-802. doi: 10.1111/j.1572-0241.2001.03874.x. PMID 11419832
- [Background] Weir MA, Fleet JL, Vinden C, Shariff SZ, Liu K, Song H, Jain AK, Gandhi S, Clark WF, Garg AX. Hyponatremia and sodium picosulfate bowel preparations in older adults. Am J Gastroenterol. 2014 May;109(5):686-94. doi: 10.1038/ajg.2014.20. Epub 2014 Mar 4. PMID 24589671
- [Background] Jin Z, Lu Y, Zhou Y, Gong B. Systematic review and meta-analysis: sodium picosulfate/magnesium citrate vs. polyethylene glycol for colonoscopy preparation. Eur J Clin Pharmacol. 2016 May;72(5):523-32. doi: 10.1007/s00228-016-2013-5. Epub 2016 Jan 28. PMID 26818765
- [Background] Maida M, Sinagra E, Morreale GC, Sferrazza S, Scalisi G, Schillaci D, Ventimiglia M, Macaluso FS, Vettori G, Conoscenti G, Di Bartolo C, Garufi S, Catarella D, Manganaro M, Virgilio CM, Camilleri S. Effectiveness of very low-volume preparation for colonoscopy: A prospective, multicenter observational study. World J Gastroenterol. 2020 Apr 28;26(16):1950-1961. doi: 10.3748/wjg.v26.i16.1950. PMID 32390705
- [Background] Halphen M, Heresbach D, Gruss HJ, Belsey J. Validation of the Harefield Cleansing Scale: a tool for the evaluation of bowel cleansing quality in both research and clinical practice. Gastrointest Endosc. 2013 Jul;78(1):121-31. doi: 10.1016/j.gie.2013.02.009. Epub 2013 Mar 24. PMID 23531426
- [Background] Lawrance IC, Willert RP, Murray K. A validated bowel-preparation tolerability questionnaire and assessment of three commonly used bowel-cleansing agents. Dig Dis Sci. 2013 Apr;58(4):926-35. doi: 10.1007/s10620-012-2449-0. Epub 2012 Oct 25. PMID 23095990
- [Background] Lyseng-Williamson KA. Macrogol (polyethylene glycol) 4000 without electrolytes in the symptomatic treatment of chronic constipation: a profile of its use. Drugs Ther Perspect. 2018;34(7):300-310. doi: 10.1007/s40267-018-0532-0. Epub 2018 Jun 15. PMID 30546252